CLINICAL TRIAL: NCT00877942
Title: Sex Differences in Early Brain Development; Brain Development in Turner Syndrome
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca Knickmeyer Santelli, Assistant Professor, University of North Carolina, Chapel Hill
Other Study IDs: K01MH083045-01 (NIH); 1K01MH083045-01 (NIH)
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For participating children with Turner Syndrome, subjects may participate in an optional blood draw for DNA extraction and hormone assays.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Typically developing children drawn from the general population
- 2: Children with Turner Syndrome

SUMMARY:
Relative risk for many psychiatric disorders differs dramatically in males and females. Early-onset disorders, such as autism, occur more often in males; other conditions, such as schizophrenia, occur at similar rates in males and females, but the sexes differ in expression. It has been hypothesized that the prevalence and expression of these disorders is related to sex differences in brain development. X-chromosome effects and early exposure to gonadal hormones are strong candidates for a causal role. The aims of the research are (1) to characterize sex differences in brain development from birth to age 2; (2) to test whether brain development is altered in infants with Turner syndrome, a well-defined genetic disorder resulting from the partial or complete loss of one of the sex chromosomes. To address aim 1, high resolution MRI, including diffusion tensor imaging (DTI), will be used to characterize sex differences in brain development from birth to age 2 in a longitudinal cohort of 250 children. To address aim 2, high resolution MRI, including DTI, will be used to compare brain development in 70 infants with Turner syndrome (X monosomy) to matched controls from aim 1. The investigators hypothesize that sex differences in gray and white matter development and in white matter maturation as assessed by DTI will be present during the first 2 years of life and that children with TS will exhibit abnormal gray and white matter development in the neonatal period.

ELIGIBILITY:
Inclusion Criteria:

* For controls a child must have a normal ultrasound at the 18 week prenatal visit and the absence of major medical or psychiatric conditions in the mother.
* Children with Turner Syndrome must have diagnosis confirmed by genetic testing.

Exclusion Criteria:

* For controls - major medical or psychiatric conditions in the mother and major medical problems or congenital conditions in the child.
* For Turner children - The study is open to all TS karyotypes except those with Y chromosome material.
* For both groups children with conditions that preclude participating in an MRI scan ( i.e. metal in the body)

Ages: 2 Weeks to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Control subjects are recruited from the Prenatal Diagnostic Clinic at UNC-Chapel Hill, which performs over 12,000 prenatal ultrasound scans a year. Please note that all pregnant women in North Carolina are referred for an ultrasound at gestational age 18 weeks as part of routine prenatal care. Subjects with Turner syndrome are identified through the UNC Turner Syndrome clinic, through advertisements with relevant local and national support groups such as the Turner Syndrome Society, and through genetic counselors and other relevant health professionals throughout the United States.
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2006-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Brain volumes on MRI | 2-4 weeks post birth

SECONDARY OUTCOMES:
Brain volumes and DTI parameters | 2-4 weeks post birth, 1 yr, 2 yr

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Knickmeyer, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States